CLINICAL TRIAL: NCT06753123
Title: Be Well at Work-Plus: A Depression and Physical Activity Intervention for Hospital Service Workers.
Brief Title: Be Well at Work-Plus: A Depression and Physical Activity Intervention for Hospital Service Workers (Aim 2)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-2024-0219; K23HL157763 (NIH)
Record Dates: First submitted 2024-12-18; First posted 2024-12-31 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Depression; Physical Inactivity
Keywords: Depression; Physical Activity; Employees; Low-income; Social needs
MeSH Terms: conditions — Depression; Sedentary Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: This is a single arm open pilot study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm: Open Pilot of Intervention (Experimental): The intervention consists of assessment of depression and work impairment, work-focused cognitive behavioral therapy, work coaching, social needs screening and referral, and text message support for mood and physical activity.
  Interventions: Behavioral: A workplace-based depression intervention for low-wage hospital workers

INTERVENTIONS:
Behavioral: A workplace-based depression intervention for low-wage hospital workers — This intervention is a remotely delivered workplace-based depression intervention that is tailored to the specific social and behavioral needs of low-wage hospital service workers. The intervention involves assessment of depression-related work impairment, work-focused cognitive behavioral therapy, work coaching, social needs screening and referral, and text message support for mood and physical activity.
  Other Names: Be Well at Work-PLUS

SUMMARY:
This study develops and tests a dynamic workplace-based depression intervention that is tailored to the specific social and behavioral needs of low-wage hospital service workers. The intervention involves assessment of depression-related work impairment, work-focused cognitive behavioral therapy, work coaching, social needs screening and referral, and text message support for mood and physical activity.

DETAILED DESCRIPTION:
Depression and physical inactivity are leading contributors to cardiometabolic diseases such as obesity, diabetes, and cardiovascular disease. Low-wage workers, who comprise one third of all workers in the U.S. and are essential to many industries, are more likely to be physically inactive and to have cardiometabolic conditions and depression, yet the participants are half as likely as higher wage workers to utilize preventive care. Targeted workplace initiatives have been successful in improving employee health, but low-wage workers are difficult to engage, in part due to a high burden of social disadvantage (e.g., food and housing insecurity, time and financial constraints). There are few, if any, workplace interventions for depression that specifically target low-wage workers and the participants unique social risk factors. This study was conceptualized using a planned adaptation approach that involves low-wage workers in the design of the intervention to increase engagement and feasibility. The study will test an evidence-based 8-session telephone-delivered depression intervention for working adults, Be Well at Work, and critical adaptations for low-wage workers: assessment and referrals for social determinants of health (e.g., food and housing insecurity, financial stress), physical activity promotion, and personalized text message behavioral support. The adapted intervention, Be Well at Work-PLUS, will be tested first in a single-arm open pilot (N=10) with exit interviews to refine the intervention content and delivery. Later, a pilot randomized controlled trial comparing Be Well at Work-PLUS to a waitlist condition (N=60) will be conducted (separate ClinicalTrials.gov study). The primary objectives are to assess acceptability, feasibility, and preliminary clinical outcomes. The primary preliminary clinical outcome is depression symptom severity, and secondary outcomes are physical activity, sleep quality, blood pressure, and BMI).

ELIGIBILITY:
Inclusion Criteria:

* part-time or full-time employment (at least 20 hours per week);
* ≥18 years old;
* employed in low-wage-earning jobs in the Environmental Services or Food & Nutrition Services Departments;
* presence of depression symptoms as measured by the Patient Health Questionnaire-9 item version; individuals who score ≥5 (indicating mild depression symptoms or higher) will be eligible;
* presence of impairment in work functioning, as measured by the Work Limitations Questionnaire; individuals who score ≥5% (indicating mild work productivity loss) will be eligible;
* possession of a cell phone with ability to receive text-messages;
* Fluent in either English or Spanish.

Exclusion Criteria:

* plan to leave Scripps employment in <6 months;
* severe mental illness or substance use condition (e.g., bipolar disorder, schizophrenia, active alcohol use disorder)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Intervention Feasibility | From enrollment to end of treatment (approximately 4 months after enrollment).
  Feasibility will be assessed by the number of intervention sessions completed. The intervention will be considered feasible if the majority of participants complete 75% (6 of 8) or more phone sessions.
Acceptability | From enrollment to end of treatment (approximately 4 months after enrollment)
  Acceptability will be assessed by the average of participants' ratings of intervention components on a 0-10 scale. Participants will rate each counseling session independently and will rate text messages on a monthly basis. The intervention will be considered acceptable if mean ratings are ≥ 7/10.

SECONDARY OUTCOMES:
Depression symptoms | From baseline through end of treatment (approximately 4 months after enrollment).
  Depression symptoms will be measured with the Patient Health Questionnaire - 9 item version (range 0-27, higher = worse depression symtpoms)
Work limitations | From baseline to end of treatment (approximately 4 months after enrollment)
  Work limitations (range: 0-100%, higher = more limitation) will be measured by the Work Limitations Questionnaire.
Perceived stress | From baseline to end of treatment (approximately 4 months after enrollment)
  Perceived stress measured by the Perceived Stress Scale (range 0-40, higher = more perceived stress).
Sleep quality | From baseline to end of treatment (approximately 4 months after enrollment)
  Sleep quality and duration as measured by the Pittsburgh Sleep Quality Index (range: 0-21, higher scores indicate worse sleep quality).
Physical activity - step count | From baseline to end of treatment (approximately 4 months after enrollment)
  Weekly step count as measured by wrist-worn FitBit watch
Body mass index (BMI) | From baseline to end of treatment (approximately 4 months after enrollment)
  A weight-to-height ratio, calculated by dividing participant's weight in kilograms by height in meters squared.
Blood pressure | From baseline to end of treatment (approximately 4 months after enrollment)
  Resting systolic and diastolic blood pressures
Physical activity - self report | From baseline to end of treatment (approximately 4 months after enrollment)
  Self-reported physical activity using the International Physical Activity Questionnaire [low/medium/high activity; metabolic equivalents (METs) per week]

CONTACTS AND LOCATIONS:
Overall Officials: Jessica L McCurley, PhD, MPH, Principal Investigator — San Diego State University
Locations (1):
- San Diego State University, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to share data as this is an open pilot study with a very small number of participants (N=10), and it would be too easy to identify individuals.